CLINICAL TRIAL: NCT00708383
Title: A Randomized Controlled Study of Human Serum Albumin and Serum Substitute Supplement as Protein Supplements for IVF Culture and the Effect on Live Birth Rates
Brief Title: in Vitro Fertilization (IVF) Media Protein and Live Birth Rates
Acronym: SSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Health Resources (Other)
Responsible Party: Marius Meintjes, Presbyterian Hospital of Dallas
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PresbyterianHDallasARTS-SSS
Record Dates: First submitted 2008-06-29; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Infertility; Pregnancy Outcome, Live Birth; In Vitro Fertilization
Keywords: embryo development; embryo quality; implantation; IVF/ICSI outcome; multiple pregnancy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Embryo culture medium supplemented with 0.5% HSA and 10% SSS
  Interventions: Other: 10% SSS embryo culture medium protein supplementation
- 2 (Active Comparator): Embryo culture medium supplemented with 0.5% HSA only
  Interventions: Other: 0.5% HSA embryo culture medium protein supplementation

INTERVENTIONS:
Other: 10% SSS embryo culture medium protein supplementation — 10% SSS in addition to the 0.5% HSA already in the culture medium.
  Arms: 1
Other: 0.5% HSA embryo culture medium protein supplementation — 0.5% HSA in the culture medium
  Arms: 2

SUMMARY:
Human conception in vivo occurs in a complex milieu that includes proteins. It has been speculated that the addition of proteins more complex than human serum albumin to culture media may improve IVF outcomes. Whether the expense, labor and risk of adding additional human-derived protein to IVF media are warranted is a question unanswered. Patients, undergoing routine IVF or ICSI, will be assigned to one of two treatment groups in a randomized, prospective clinical trial . Embryos will be cultured in either media supplemented with human serum albumin (HSA) as a solitary protein supplement or in media supplemented with HSA + SSS from the 2-PN stage until the time of embryo transfer. Clinical endpoints monitored will be implantation rate, clinical pregnancy rate and live birth rate. It is expected that the supplementation of commercial embryo culture media containing HSA with the more complex protein source, SSS, will result in an overall increase in implantation, clinical pregnancy, and live birth rates. In the balance, protein enrichment of media may represent opportunities to simultaneously increase the live birth rate and reduce the incidence of multiple gestations.

DETAILED DESCRIPTION:
Purpose: The purpose of this comparison is to determine the best of two protein sources in the embryo culture media for future use in the Presbyterian Assisted Reproductive Technology Services (ARTS) Program.

Background: For embryos to grow in the incubator, a protein source is essential in the embryo culture media. Currently, HSA (simple protein) is used as the sole protein source in the embryo culture media of the Presbyterian ARTS laboratories. Literature suggests that by adding globulins, e.g. SSS (increasing the complexity of the protein source) to the culture media, the resultant embryos may be of better quality and have an increased chance to produce a pregnancy. HSA and/or SSS are routinely used as a standard protein source by most commercial human IVF programs. Both sources of proteins are FDA approved for use in human embryo culture media. The goal is to switch to the better protein source (existing HSA vs. more complex SSS), without compromising established pregnancy rates. To do this responsibly, Presbyterian ARTS Program feels that it should introduce the potential improved formulation (existing culture media supplemented with SSS) by comparing it in a randomized, prospective way with the existing culture system (existing culture media supplemented with HSA).

Project Summary: Study design: The study will be conducted in a prospective, randomized way. Two treatment groups are considered: 1) culture media supplemented with HSA 2) Culture media supplemented with SSS. To allow for the well-documented decline in pregnancy rates with increased age, patients will be randomized within 4 age groups and 7 physicians within each treatment (blocked for age and physician within treatments). The age groups are: donor eggs; <35 years; 35 to 37 years; and 38 to 40 years as determined on the day of egg retrieval.

Endpoints Measured: The endpoints measured will be embryo cryopreservation-biochemical pregnancy-, clinical pregnancy-, ongoing pregnancy-, live birth- and embryo implantation rates.

Number of Patients in the Study: To detect a difference of 10% in pregnancy rates, 150 patients should be included in each treatment group. With the current patient volume, it should take less than one year to complete the study. Differences in implantation rates may be detected earlier (more embryos transferred than patients enrolled). Should significance differences in pregnancy rates become evident before the full number of patients is enrolled, the study may be terminated.

Study Location: The study will be conducted simultaneously at both ARTS facilities of Presbyterian Hospital of Dallas and Presbyterian Hospital of Plano.

Criteria for Inclusion of Subjects: All patients undergoing a first IVF cycle or any donor oocyte cycle is eligible to participate in this laboratory comparison. The eggs may be fertilized with conventional IVF methodology or by using intracytoplasmic sperm injection (ICSI). When performing ICSI, ejaculated sperm must be used. Patients using their own eggs must be 40 years of age or younger on the day of egg retrieval. The Presbyterian Hospital ARTS Program performed ~900 commercial egg retrievals in 2000. Of these, ~500 would have met the inclusion criteria of this study.

Criteria for Exclusion of Subjects: To reduce the tremendous patient variability seen in the infertile patient population, only first cycle patients 40 years of age or younger on the day of egg retrieval should participate.

Sources of Research Material: Patients will be enrolled in this study from the regular patient pool presented to the Presbyterian ARTS Program for treatment of infertility. Data will not be collected specifically for research purposes. Data to be used are collected on all ARTS patients, regardless of participation in the study.

Recruitment of Subjects: Subjects for this study will be recruited from the regular patient pool presented to the ARTS Program for the treatment of infertility. Patients that will meet the inclusion criteria of this study can be identified prospectively. Information about the study will be included in the routine, biweekly, group laboratory and nursing orientation sessions. Patients meeting the inclusion criteria for the study will be presented with the study consent along with their regular IVF consents and asked to consider joining the study. The attending physician, the physician's nurse, the ARTS Scientific Director, attending embryologist or ARTS nurse may approach these patients.

Potential Risks: Patients consenting to the comparison will allow their embryos to be cultured in either the standard HSA-supplemented embryo culture media or in embryo culture media supplemented with SSS. HSA-supplemented culture media is the current standard in this program. SSS-supplemented media is used routinely in many other commercial IVF-programs and for cryopreservation of embryos in the Presbyterian ARTS Program. Both HSA and SSS is FDA approved for use in human embryo culture media. Culture conditions and ingredients that will be applied are not experimental. The embryos will not be exposed to procedures or substances considered not being industry standard in human IVF laboratories. To the best knowledge of Presbyterian Hospital ARTS Program, published literature suggests that the SSS-supplemented culture media may do better rather than worse under the conditions proposed for this study. However, when HSA and SSS are compared in a controlled, randomized way as suggested in this comparison, the ARTS Program can not guarantee that the pregnancy outcome will be equivalent for both treatment groups (HSA vs. SSS). Therefore, by being randomized, a patient may be included in a group with a lower success rate.

Special Precautions: If it should become clear early in the study that the SSS treatment outcome is inferior to the current culture system (HSA) in place, the study will be discontinued.

Procedures to Maintain Confidentiality: No additional information will be collected from study patients than that not otherwise collected from ARTS patients. Data collected will be treated in the same way as for other ARTS patients. The ARTS Scientific Director, aided by 6 embryologists will keep record of the number of patients enrolled in the study, randomization procedures, treatment allocations and outcome of the endpoints measured by treatment. Nursing and administrative personnel will not have access to the treatment-specific data. The treatment allocation sheets will be kept in the two IVF laboratories. Only the embryologists have access to these laboratories. The executed consent forms will be treated like all other consents pertaining to the IVF cycle and be filed in the patient's chart in the consent section. Copies will only be made for the patients.

Potential Benefits: The patients directly involved in this study may benefit if their treatment-group provide higher pregnancy rates than the current standard treatment protocol (HSA only). For future ARTS patients, information obtained from this study may determine the better protein source or the equivalency of both protein sources for use in culture media in the ARTS laboratory to allow the best possible pregnancy rates. Only a very few programs have the patient volume and ability to examine this in a controlled manner.

Risk/Benefit Assessment: The proteins to be compared are both FDA approved for use in human embryo culture media. Furthermore, industry-standard culture conditions and methodology will be used throughout the study period. Literature suggests that the embryo quality and pregnancy outcome should improve rather than deteriorate when increasing the complexity of the protein source. The Presbyterian ARTS Program perceives the risk to be minimal. This is a responsible way of introducing a new variable with potential benefits into the ARTS IVF laboratory without risking the established, successful embryo culture protocol. By not constantly seeking ways to improve the pregnancy rates for our patients, Presbyterian ARTS Program runs the risk of becoming a stagnant, outdated IVF program. The ability to compare these variables (protein source) in a randomized, prospective way will be invaluable to the ARTS community in general. The researchers can not guarantee that the outcomes for all treatment groups will be equivalent. Therefore, it is possible that a patient may be included in a treatment group with a lower success rate.

ELIGIBILITY:
Inclusion Criteria:

* First IVF or any donor oocyte cycle
* The eggs may be fertilized with conventional IVF methodology or by using intracytoplasmic sperm injection (ICSI).
* When performing ICSI, ejaculated sperm must be used
* 40 years of age or younger on the day of egg retrieval

Exclusion Criteria:

* One or more previous failed IVF cycles
* Use of epididymal or testicular sperm for ICSI
* Older than 40 years of age

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 538 (Actual)
Dates: Start 2001-09; Primary Completion 2002-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Live birth | 9 months

SECONDARY OUTCOMES:
Implantation rate | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marius Meintjes, PhD, Principal Investigator — Texas Health Resources
Locations (2):
- United States (2):
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Presbyterian Hospital of Plano, Plano, Texas

REFERENCES:
- [Derived] Meintjes M, Chantilis SJ, Ward DC, Douglas JD, Rodriguez AJ, Guerami AR, Bookout DM, Barnett BD, Madden JD. A randomized controlled study of human serum albumin and serum substitute supplement as protein supplements for IVF culture and the effect on live birth rates. Hum Reprod. 2009 Apr;24(4):782-9. doi: 10.1093/humrep/den396. Epub 2009 Jan 14. PMID 19147504